CLINICAL TRIAL: NCT07331025
Title: Ultrasound Detection of Early Facial Muscle Changes in FSHD: Thickness and Echo Intensity Findings - A Cross-Sectional Comparison With Healthy Adults
Brief Title: Ultrasound Detection of Early Facial Muscle Changes in FSHD: Thickness and Echo Intensity Findings
Acronym: FACIAL-FSHD
Status: Completed | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Havvanur Albayrak, Physical Medicine and Rehabilitation Specialist, Koç University
Other Study IDs: 2023.278.IRB1.092; 2023.278.IRB1.092 (Other: Koç University Institutional Review Board)
Record Dates: First submitted 2025-12-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Facioscapulohumeral Muscular Dystrophy; Facioscapulohumeral Muscular Dystrophy 1; Neuromuscular Disease
Keywords: facioscapulohumeral muscular dystrophy; facial muscles; muscle ultrasound; muscle echogenicity; muscle thickness; imaging biomarker
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FSHD patients: Individuals with genetically confirmed facioscapulohumeral muscular dystrophy type 1 who underwent bilateral facial muscle ultrasound assessment. No intervention was applied.
- Healthy Controls: Age- and sex-matched healthy volunteers without neuromuscular disease.

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is characterized by early and significant involvement of facial muscles; however, objective imaging data focusing on facial muscles are limited. Facial ultrasound can serve as a sensitive imaging biomarker and outcome measure by capturing regional structural changes in facial muscles associated with disease progression in FSHD patients.

The aim of this study is to compare facial muscle thickness and echo density between FSHD patients and healthy controls using ultrasound and to examine the relationships between ultrasound findings and clinical parameters.

This study will include 20 patients with genetically confirmed FSHD1 diagnosis and 19 age- and sex-matched healthy controls. Using musculoskeletal ultrasound, bilateral evaluation of selected facial muscles (Orbicularis oculi, orbicularis oris, zygomaticus major, and buccinator) will be performed by two different researchers, and muscle thickness and muscle echo density will be recorded. Inter-rater reliability will be assessed using intraclass correlation coefficients. Group comparisons and correlation analyses will be performed with clinical scores, symptom duration, and D4Z4 repeat size.

The results will evaluate whether ultrasound can reliably detect structural changes in FSHD that cannot be captured by traditional clinical assessments, and if significant, will suggest that ultrasound can serve as a sensitive imaging biomarker for early and region-specific facial muscle involvement in FSHD.

DETAILED DESCRIPTION:
Facioscapulohumeral muscular dystrophy (FSHD) is a hereditary neuromuscular disorder characterized by progressive muscle weakness, showing early and significant involvement of facial muscles. Despite their diagnostic and functional importance, facial muscles are often underrepresented in imaging-based assessments of disease involvement. This observational, cross-sectional study was designed to compare structural changes in selected facial muscles of individuals with genetically confirmed FSHD with healthy controls using musculoskeletal ultrasound. The study focuses on the quantitative assessment of muscle thickness and the qualitative assessment of muscle echo density as indicators of atrophy and fat infiltration. Bilateral ultrasound examinations will be performed on facial muscles, including the orbicularis oculi, orbicularis oris, zygomaticus major, and buccinator muscles, which play a role in facial expression and oral function. Imaging findings will be evaluated in relation to clinical features to investigate whether facial muscle ultrasound can provide region-specific information not captured by global disease severity scores. This study aims to characterize facial muscle involvement using a non-invasive and accessible imaging method, contribute to the understanding of early and subclinical facial muscle changes in FSHD, and support the potential role of ultrasound as an imaging biomarker in neuromuscular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 years
* Genetically confirmed facioscapulohumeral muscular dystrophy type 1 (FSHD1) (patient group)
* Age- and sex-matched healthy volunteers without neuromuscular disease (control group)
* Ability to provide written informed consent

Exclusion Criteria:

* Presence of other neurological or neuromuscular disorders
* History of facial palsy or facial trauma
* Botulinum toxin injection to facial muscles within the last 6 months
* Inability to cooperate with ultrasound assessment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of adults with genetically confirmed facioscapulohumeral muscular dystrophy type 1 and age- and sex-matched healthy volunteers. Participants were recruited from a tertiary neuromuscular disease center and underwent a single-session bilateral facial muscle ultrasound assessment.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Facial muscle thickness measured by ultrasound | Baseline
  Bilateral thickness (in millimeters) of the orbicularis oculi, orbicularis oris (superficial and deep layers), zygomaticus major, and buccinator muscles measured using B-mode musculoskeletal ultrasound at standardized anatomical reference points.
Facial muscle echo intensity | Baseline
  Muscle echogenicity of the same facial muscles assessed bilaterally using the Modified Heckmatt Scale (grades 1-4) to evaluate structural changes and fatty infiltration on B-mode ultrasound images.

SECONDARY OUTCOMES:
Inter-rater reliability of facial muscle ultrasound measurements | Baseline
  Agreement between independent raters assessed using intraclass correlation coefficients for facial muscle thickness and echo intensity measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Havvanur Albayrak, Principal Investigator — Koç University School of Medicine
Locations (1):
- Koç University Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size, the rare disease nature of the study population, and the potential risk of participant re-identification. In addition, specific informed consent for public data sharing was not obtained.